CLINICAL TRIAL: NCT07097753
Title: A Retrospective Cohort Before-After Study Comparing the Prognostic Outcomes of MIPPED-C With Open Surgical Necrosectomy in Infected Pancreatic Necrosis
Brief Title: Comparison of MIPPED-C and Surgical Necrosectomy in Pancreatic Necrosis Outcomes
Status: Enrolling by invitation | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20250529075134604
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-05

CONDITIONS: Acute Pancreatitis (AP); Acute Pancreatitis With Infected Necrosis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Open surgical debridement of necrotic tissue
- Minimally Invasive Partitioned Pancreatic Debridement and Enhanced Cross-Drainage

SUMMARY:
This study is a retrospective, single-center, pre-post controlled clinical study. Patients (n=48) who underwent the MIPPED-C surgical procedure after January 1, 2019 were designated as the treatment group. Patients who were admitted to the hospital from January 1, 2014 to December 31, 2018 and underwent traditional open surgery were retrospectively evaluated by surgeons, radiologists, and interventionalists, and then matched for propensity score with a 1:2 ratio. 96 patients who underwent traditional open surgery were selected as the control group. The treatment group underwent the MIPPED-C surgery, while the control group underwent the traditional open necrotic tissue debridement procedure. The differences in inflammatory indicators, SIRS response, immune indicators, organ function indicators, and imaging changes of the two groups of patients at the time of admission, before the operation, and after the operation were retrospectively collected. The survival status, postoperative complications, re-intervention status, hospital stay, ICU stay, and hospitalization costs of the two groups of patients after the operation were also collected.

ELIGIBILITY:
Inclusion Criteria:(1) age ≥18 years; (2) a confirmed diagnosis of infected pancreatic necrosis (IPN) based on imaging (e.g., presence of gas within necrosis) and clinical indicators (e.g., fever, leukocytosis, or positive cultures); (3) underwent either the MIPPED-C procedure or OSN as the definitive surgical intervention; and (4) had a minimum follow-up period of 90 days postoperatively.

Exclusion Criteria:(1) non-infected pancreatic necrosis; (2) receipt of interventions other than MIPPED-C or OSN (e.g., endoscopic or purely percutaneous approaches); (3) prior history of IPN surgery or other major abdominal surgery that could confound surgical outcomes; or (4) incomplete follow-up data or loss to follow-up within 90 days after surgery.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent traditional pancreatic debridement surgery and MIPPED-C IPN at Ruijin Hospital, affiliated to Shanghai Jiao Tong University School of Medicine from January 1, 2014 to December 31, 2023
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | Half a year after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Department of Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided